CLINICAL TRIAL: NCT03987191
Title: Successful Transition From Insulin Pump to Multiple Daily Injections Using Insulin Degludec in Adults With Type 1 Diabetes
Brief Title: Insulin Pump to Multiple Daily Injection Transition Clinical Trial
Acronym: TRANSITION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-0924
Record Dates: First submitted 2019-06-05; First posted 2019-06-14 (Actual); Results first posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care Transition (Active Comparator): Stopping of insulin pump on the day of randomization and starting insulin degludec in 1:1 ratio (same units as total basal insulin on pump) and insulin Aspart for meals and corrections
  Interventions: Drug: Multiple daily ijnection using Insulin Degludec and Insulin Aspart
- Inverstigational Transition (Experimental): Administration of insulin degludec in 1:1 ratio (same units as total basal insulin on pump) on the day of randomization AND concomitant use of the insulin pump for 48 hours from transition, where insulin pump basal rate will be reduced by 50% during the first 24 hours from transition and by 75% during 24 to 48 hours from transition. Insulin pump will be disconnected after 48 hours from transition
  Interventions: Drug: Multiple daily ijnection using Insulin Degludec and Insulin Aspart

INTERVENTIONS:
Drug: Multiple daily ijnection using Insulin Degludec and Insulin Aspart — Drug: Insulin Degludec and insulin Aspart Pharmaceutical form: Solution for injection Route of administration: Subcutaneous

SUMMARY:
This randomized controlled, two arms, investigator initiated, intervention study is aimed to examine an investigational approach in contrast to the clinical standard of 1:1 dose basal insulin conversion in an attempt to lower the incidence and/or duration of hyperglycemia after transition from insulin pump to multiple daily injections in adults with type 1 diabetes.

DETAILED DESCRIPTION:
Second generation long acting insulin, insulin degludec, has been shown to improve glycemic control and reduce hypoglycemia in patients with type 1 diabetes and insulin treated type 2 diabetes. However, it takes about 48 hours before glycemic benefits are noticeable. Therefore, transition from insulin pump to multiple daily injection using insulin degludec is associated with hyperglycemia during first 48 hours of transition. Considering this, this study proposes to evaluate an investigational strategy to improve glycemic control during transition from insulin pump to multiple daily injections using insulin degludec and insulin aspart.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤ 65 years
2. Patients with T1D diagnosed for at least 12 months
3. Point-of-care HbA1c levels between ≥6.5% and ≤ 8.5%
4. Patients on CSII (any insulin pump) for at least past 6 months
5. Willing and able to wear a blinded CGM during the time of study period
6. Willing to perform self-monitoring of blood glucose (SMBG) at least 4 times a day
7. Ability to provide informed consent before any trial-related activities
8. Not willing to or plan any travel out of Colorado during the 3 weeks of study period
9. Willing to use insulin degludec in the morning once a day

Exclusion Criteria:

1. Age <18 years and > 65years
2. HbA1c >8.5 % at screening
3. Less than 12 months of insulin treatment
4. Patients on 670G or Tandem Control IQ (Medtronic and Tandem Hybrid Closed-loop systems) and not willing use manual mode during the study period
5. Patients with T1D using any glucose lowering medications other than insulin
6. Pregnancy, breast feeding, and positive pregnancy test during screening
7. Women of childbearing age wanting to become pregnant or not using adequate contraceptive measures
8. Current or recent (< 2 weeks prior to visit 1) use of any steroidal medication, or anticipated steroidal treatment, during the study period
9. eGFR below 45 ml/min/1.73 m^2 using MDRD formula
10. History of severe hypoglycemia in the previous 3 months
11. History of diabetic ketoacidosis (DKA) requiring hospitalization in the past 3 months
12. History of allergy to any form of insulin or its excipients
13. History of allergy to adhesives
14. Unwilling to use blinded CGM during the study period
15. Unwilling to perform SMPG at least 4 times a day
16. Known history of alcohol abuse or illicit drug use within 6 months prior to screening
17. Use of investigational drugs within 5 half-lives prior to screening
18. Participation to other study trials during the study period
19. Elevated liver enzymes (AST and ALT) 3 times the upper limit of normal
20. Hypoglycemia unawareness defined as GOLD score ≥4 [20]
21. Any comorbidities or medical conditions that make a person unfit for the study at the discretion of the investigators
22. Anticipated travel across different time zones (difference greater than 4 hours) or anticipated change in physical activities or diet at the discretion of the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Viral Shah, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Barbara Davis Center for Diabetes, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified academic researchers may request access to de-identified participant level data related to the study. The request letter with details such as reasons for data request, plan for data analysis, publication and so on should be emailed/mailed to the PI of the study (viral.shah@cuanschutz.edu).
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after the publication. The data sharing details will be provided in the manuscript.
Access Criteria: The committee (PI, statistician and Sponsor) will decide on appropriate request for data sharing.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 screen failed, 1 participant was lost to follow-up prior to screening, and 2 withdrew from study prior to randomization.
Groups:
- Investigational Transition: Administration of insulin degludec in 1:1 ratio (same units as total basal insulin on pump) on the day of randomization AND concomitant use of the insulin pump for 48 hours from transition, where insulin pump basal rate will be reduced by 50% during the first 24 hours from transition and by 75% during 24 to 48 hours from transition. Insulin pump will be disconnected after 48 hours from transition
  Multiple daily ijnection using Insulin Degludec and Insulin Aspart: Drug: Insulin Degludec and insulin Aspart Pharmaceutical form: Solution for injection Route of administration: Subcutaneous
Period: Overall Study
Arm/Group | Standard of Care Transition | Investigational Transition
Started | 17 | 15
Data Collected | 17 | 13
Completed | 17 | 13
Not Completed | 0 | 2
Not completed — COVID-19 related research disruption | 0 | 2

BASELINE CHARACTERISTICS:
Population: No data is available for the two participants who did not have data collected due to COVID-19-related research disruption.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Transition | Investigational Transition | Total
Number analyzed (Participants) | 17 | 13 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.7 (9.1) | 38.2 (9.5) | 36.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 8 | 7 | 15
Race/Ethnicity, Customized [Number; unit: Number of participants]
  White | 15 | 13 | 28
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 17 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: Time Spent With CGM Glucose Levels >180mg/dl Between Two Groups
Description: The primary outcome will be time spent in CGM glucose >180 mg/dL (hyperglycemia) during 7days of randomization period between two groups.
Time Frame: 7 days from the randomization
Measure: Median (Inter-Quartile Range); unit: percentage of time spent >180 mg/dL
Arm/Group | Standard of Care Transition | Investigational Transition
Number analyzed (Participants) | 17 | 13
percentage of time spent >180 mg/dL | 46.3 [43.5 to 49.1] | 38.5 [30.7 to 47.1]

2. Secondary Outcome: Time Spent in CGM-measured "Time-in-range"(Glucose Levels ≥70 mg /dl and ≤180 mg/dl) Between Two Groups
Description: CGM TIR between two groups
Time Frame: 7 days from the randomization
Measure: Median (Inter-Quartile Range); unit: percentage of time spent in range
Arm/Group | Standard of Care Transition | Investigational Transition
Number analyzed (Participants) | 17 | 13
percentage of time spent in range | 47.8 [44.1 to 52.1] | 56.5 [51.0 to 63.9]

3. Secondary Outcome: Time Spent in CGM-measured Hypoglycemia < 70 mg/dl Between Two Groups
Description: CGM time below 70 between two groups
Time Frame: 7 days from the randomization
Measure: Median (Inter-Quartile Range); unit: percentage of time below range
Arm/Group | Standard of Care Transition | Investigational Transition
Number analyzed (Participants) | 17 | 13
percentage of time below range | 3.9 [2.4 to 7.2] | 2.1 [1.0 to 5.4]

4. Secondary Outcome: Number of Participants With Severe Hypoglycemia as Defined by the ADA (Severe Cognitive Impairment Requiring External Assistance for Recovery) and Severe Hyperglycemia (BG≥250 Needing Hospitalization) Between Two Groups
Description: Frequency of SH and DKA between two groups
Time Frame: 7 days from the randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Transition | Investigational Transition
Number analyzed (Participants) | 17 | 13
Participants
  Participants with Severe Hypoglycemia | 0 | 0
  Participants with Diabetic Ketoacidosis | 0 | 0

5. Secondary Outcome: Number of Boluses (Correction Boluses) Between Groups During First 72 Hours of Randomization
Description: no of correction boluses between two groups
Time Frame: 72 hours from the randomization
Measure: Median (Inter-Quartile Range); unit: Boluses per day
Arm/Group | Standard of Care Transition | Investigational Transition
Number analyzed (Participants) | 17 | 13
Boluses per day | 6.5 [4.5 to 8.7] | 4.0 [3.0 to 6.5]

6. Secondary Outcome: Insulin Delivery Satisfaction (IDSS Survey) Between Two Groups
Description: PRO between two groups. The Insulin delivery satisfaction survey (IDSS) measures diabetes patients' satisfaction with their insulin delivery system. Possible scores range from 1-5, with higher scores indicating higher satisfaction and a better outcome.
Time Frame: 7 days from the randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care Transition | Investigational Transition
Number analyzed (Participants) | 17 | 13
score on a scale | 3.9 [3.9 to 4.3] | 3.9 [3.8 to 4.1]

7. Secondary Outcome: Work Productivity and Activity Impairment (WPAI:SHP Version 2 Questionnaire) Between Two Groups
Description: PRO between two groups
Time Frame: 7 days from the randomization
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | Standard of Care Transition | Investigational Transition
Number analyzed (Participants) | 17 | 13
Percent
  Percent work time missed due to problem | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Percent impairment while working | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  Percent overall work impairment | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Percent activity impairment due to problem | 0.1 [0.1 to 0.2] | 0.2 [0.2 to 0.4]

ADVERSE EVENTS:
Time Frame: 7 Days
Arm/Group | Standard of Care Transition | Investigational Transition
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/13
Other Adverse Events (participants affected / at risk) | 0/17 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Transition (N=17) | Investigational Transition (N=13)
AE unrelated to the study (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Common cold

LIMITATIONS AND CAVEATS:
Single Center study with small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/91/NCT03987191/Prot_SAP_000.pdf